CLINICAL TRIAL: NCT01796769
Title: Multidisciplinary and Coordinated Follow-up Based on a Telemonitoring Web Platform for Improving Continuous Positive Airway Pressure (CPAP) Compliance in Low Cardiovascular Risk Sleep Apnea Patients
Brief Title: Multidisciplinary and Coordinated Follow-up Based on a Telemonitoring Web Platform for Improving CPAP Compliance in Low Cardiovascular Risk Sleep Apnea Patients : OPTISAS 1 Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fédération Française de Pneumologie (Other)
Collaborators: Federation of Medical Specialties (Other)
Responsible Party: Principal Investigator, Jean Louis PEPIN, Professor, PhD, Hospital Grenoble France, Fédération Française de Pneumologie
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-FFPO-01
Record Dates: First submitted 2013-02-15; First posted 2013-02-22 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Sleep Apnea Syndrome; Low Cardiovascular Risk
Keywords: Obstructive Sleep Apnea Syndrome; Telemedicine; Patient Compliance
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Patient Compliance | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Experimental)
  Interventions: Device: Continuous Positive Airway Pressure (CPAP) in sleep apnea patients
- Telemedicine (Active Comparator)
  Interventions: Device: Continuous Positive Airway Pressure (CPAP) in sleep apnea patients

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) in sleep apnea patients — Usual CPAP treatment in sleep apnea patients
  Arms: Conventional
Device: Continuous Positive Airway Pressure (CPAP) in sleep apnea patients — CPAP treatment with telemedicine system
  Arms: Telemedicine

SUMMARY:
Targeted population:

Sleep apnea patients at low cardiovascular risk newly treated by CPAP

Hypothesis:

Six months CPAP compliance might be greater in the telemonitoring arm compared to usual CPAP care.

Main goal:

To compare 6-months CPAP compliance when Sleep Apnea patients at low cardiovascular risk are randomly allocated to usual CPAP care or a multidisciplinary and coordinated follow-up based on a telemonitoring web platform.

DETAILED DESCRIPTION:
Study procedures:

The telemonitoring system will involve respiratory physicians, home care providers and include regular assessments of oximetry, CPAP compliance, side effects and residual events.

Secured data transmission to medical staff computers and secured websites will allow easy telemonitoring. Automatic algorithms have been built-up for early adjustment of CPAP treatment in case of side effects, leaks and persistent residual events.

An interim analysis will be performed when 200 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 78 years
* Men and women
* AHI > 30 / hour
* Patient with low cardiovascular score (<5% defined by European SCORE)
* Patient affiliated to the national health insurance
* Willingness to use a telemonitoring system

Exclusion Criteria:

* Known cardiovascular disease (i.e. transient ischemic attack, stroke, coronary artery disease)
* Central sleep apnea syndrome
* Previous CPAP treatment with respiratory support for sleep respiratory trouble
* Cardiac failure
* Hypercapnic chronic respiratory failure (daytime PaCO2 > 50 mmHg)
* Terminal disease

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 936 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline CPAP compliance at 6 months | day 0 and month 6
  CPAP compliance evolution by comparing baseline and 6 months measurements. CPAP compliance is assessed at month 6 in the two groups.

SECONDARY OUTCOMES:
Subjective Sleepiness | inclusion and month 6
  Sleepiness is assessed with Epworth Sleepiness Scale at inclusion and month 6 in the two groups
Fatigue | inclusion and month 6
  Fatigue is assessed with Pichot Scale at inclusion and month 6 in the two groups
Quality of Life | inclusion and month 6
  Quality of life is assessed with SF-12 questionnaire at inclusion and month 6 in the two groups
Health status | inclusion and month 6
  Health status is assessed with EQ-5D questionnaire at inclusion and month 6 in the two groups
Cost analysis | month 6
  Cost analysis will include all key resources associated with the telemonitoring intervention and related health (referrals, consultations, resource use)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis PEPIN, Prof, PhD, Principal Investigator — Functional Cardio-Respiratory Exploration Laboratory - University Hospital Grenoble - France
Locations (32):
- France (32):
  - Respiratory physician in private practice, Albertville
  - Respiratory physician in private practice, Annecy
  - Respiratory physician in private practice, Bordeaux
  - General Hospital, Cannes
  - General Hospital, Denain
  - Dieulefit Santé Clinic, Dieulefit
  - Respiratory physician in private practice, Échirolles
  - Saint Vincent Clinic, Épernay
  - University Hospital, Grenoble
  - Respiratory physician in private practice, Grenoble
  - Respiratory physician in private practice, La Rochelle
  - University Hospital Calmette, Lille
  - La Louvière Clinic, Lille
  - General Hospital, Magny-en-Vexin
  - Ambroise Paré Hospital, Marseille
  - General Hospital, Montélimar
  - Respiratory physician in private practice, Montigny-lès-Metz
  - Respiratory physician in private practice, Nîmes
  - Les Rieux Clinic, Nyons
  - Hospital Bichat Claude Bernard, Paris
  - Respiratory physician in private practice, Reims
  - University Hospital, Rouen
  - General Hospital, Saint-Avold
  - Respiratory physician in private practice, Saint-Etienne
  - Respiratory physician in private practice, Saint-Ismier
  - Respiratory physician in private practice, Saint-Laurent-du-Var
  - Respiratory physician in private practice, Saint-Omer
  - Respiratory physician in private practice, Six-Fours-les-Plages
  - Respiratory physician in private practice, Toulon
  - Respiratory physician in private practice, Valence
  - Tessier Clinic, Valenciennes
  - Hospital Nord Ouest, Villefranche-sur-Saône